CLINICAL TRIAL: NCT05723341
Title: Comparison of Postoperative Analgesic Effects of Ultrasonography-Guided Paravertebral Block and Subcostal Transversus Abdominis Plane Block in Patients Undergoing Laparoscopic Nephrectomy
Brief Title: Comparison of Paravertebral Block and Subcostal Transversus Abdominis Plane Block in Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1276671
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Analgesia; Anesthesia; Pain, Postoperative
Keywords: Paravertebral Block; Subcostal Transversus Abdominis Plane Block; Postoperative Controlled Analgesia; Postoperative Pain; Laparoscopic Nephrectomy
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Intervention Model Description: RANDOMISED SINGLE BLINDED INTERVENTIONAL
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paravertebral Block Group (Active Comparator): In this group, preoperative ultrasound-guided paravertebral block will be performed ipsilateraly via peripheral block needle with 20 ml bupivacaine %0,25 in the paravertebral space.
  Interventions: Drug: Bupivacain; Drug: Morphine
- Subcostal Transversus Abdominis Plane Block Group (Active Comparator): In this group, preoperative ultrasound-guided subcostal transversus abdominis plane block will be performed ipsilateraly via peripheral block needle with 20 ml bupivacaine %0,25 into the fascial plane between erector spine muscle and transverse process
  Interventions: Drug: Bupivacain; Drug: Morphine
- Intravenous Patient Controlled Analgesia (Active Comparator): In this group, postoperative patient controlled analgesia with morphine will be preferred for postoperative analgesia method.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Bupivacain — %0,25
  Other Names: Marcaine
  Arms: Paravertebral Block Group; Subcostal Transversus Abdominis Plane Block Group
Drug: Morphine — In this group, patients will be postoperatively administered patient-controlled analgesia with morphine only.
  Other Names: Morphine Sulfate

SUMMARY:
Most of the patients undergoing laparoscopic partial/radical nephrectomy can experience moderate or severe postoperative pain, and inadequate control of this pain can cause negative consequences such as development of chronic pain, pulmonary and cardiac events, and side effects of long term opioid usage. Due to these adverse outcomes, ultrasonography-guided plane blocks can be beneficial for these patients to decrease opioid consumption. In this study, the investigators aim to compare ultrasonography-guided plane blocks: Paravertebral block and subcostal transversus abdominis plane block and traditional method: patient controlled analgesia with opioids. The investigators hypothesized that analgesic efficacy in both paravertebral and subcostal TAP blocks will have similar outcomes but better than traditional method.

DETAILED DESCRIPTION:
More than half of patients undergoing laparoscopic partial/radical nephrectomy develop moderate or severe postoperative pain. Inadequate control of postoperative pain may delay early mobilization and rehabilitation, increase pulmonary and thromboembolic events, prolong hospital stay, and decrease patient satisfaction. Inadequate postoperative pain control may lead to the development of chronic pain, resulting in long-term opioid use. In the traditional analgesia model provided with opioids, patients may develop side effects such as nausea, vomiting, hypotension, loss of consciousness, and respiratory depression. For this reason, it would be more rational to provide analgesia with regional methods, which are decided according to the suitability of the patient and the surgical procedure, rather than the use of intravenous drugs. Ultrasonography-guided plane blocks, one of the main elements of multimodal analgesia, are used more frequently with the introduction of ultrasonography into daily practice. These blocks are frequently preferred in daily practice as they reduce opioid consumption by providing effective postoperative analgesia with low complication rates and ease of application.

In the ultrasonography-guided paravertebral block, local anesthetic is injected into the triangle constituted by superior costotransvers ligament, parietal pleura and vertebral body where the spinal nerves emerge from the intervertebral foramen. Ipsilateral somatic and sympathetic nerve blockade is observed. It is a body block that can be used to provide both analgesia and anesthesia. Paravertebral block provides successful postoperative analgesia, reduces the decline in postoperative respiratory function, accelerates the recovery of respiratory mechanics, and reduces postoperative vomiting, allowing earlier initiation of oral intake.

Ultrasonography-guided subcostal transversus abdominis plane block is a relatively safe and simple body block in which local anesthetic is injected into the fascial plane located between posterior rectus sheath and transversus abdominis muscle. The transversus abdominis plane is the fascial plane superficial to the transversus abdominis muscle, the innermost muscular layer of the anterolateral abdominal wall. The subcostal transversus abdominis plane block ideally anesthetizes the intercostal nerves T6-T9 between the rectus abdominis sheath and the transversus abdominis muscle. It is a truncal block that has drawn attention recently, both because it is easier to apply and because it is a more peripheral block.

In this study the investigators aim to compare the effects of two truncal blocks on postoperative pain, morphine consumption, chronic pain and complications.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75
* Patients who are ASA (American Society of Anesthesiology): I-II
* Patients who will have laparoscopic partial/radical nephrectomy
* Patients who volunteer to participate in the study

Exclusion Criteria:

* Patients with any kind of coagulopathy
* Patients with severe cardiac, pulmonary, renal or liver disease
* Patients who have difficulty comprehending the IV PCA device
* Patients with local anesthetic allergy
* Patients with chronic opioid use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Intravenous Total Morphine Consumption | Up to 24 hours
  The total dosage of intravenous morphine consumption in 24 hours.

SECONDARY OUTCOMES:
Postoperative Visual Analog Score (VAS) | Up to 24 hours
  A visual analog score (VAS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Rescue analgesia administration amounts | Up to 24 hours
  Time of postoperative rescue analgesic requirement time.
Incidence of complications due to the regional blocks | Up to first week
  Incidence of hematoma, pneumothorax (pleural puncture), local anesthetic toxicity, infection vs.
Chronic postoperative pain | Up to 90th day
  Patients' chronic pain will be assessed by the examiner questioning each patient about the pain status on postoperative 90th day.
Lenght of Hospital Stay | Up to first week
  Lenght of Hospital Stay

OTHER OUTCOMES:
Indidence of PONV (postoperative nausea and vomiting) | Up to 24 hours
  Incidence of postoperative nausea and vomiting
Respiratuar Depression | Up to 24 hours
  Incidence of respiratory depression due to iv orphine in the postoperative follow-up.
Postoperative Ramsay Sedation Scale (RSS) | Up to 24 hours
  Ramsay sedation scale requires the patient to rate their sedation on a defined scale. For example, 1: anxious and agitated or restless, or both 2: cooperative, oriented and tranquil 3: responds to commands only 4: brisk response to stimulus 5: sluggish response to stimulus 6: no response to stimulus.
Itching | Up to 24 hours
  Incidence of itching due to iv morphine in the postoperative follow-up.
Surgeon Satisfaction | Up to 24 hours
  Satisfaction score, 0: very unsatisfied 3: very unsatisfied.
Patient Satisfaction | Up to 24 hours
  Satisfaction score, 0: very unsatisfied 3: very unsatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, MD, Principal Investigator — Istanbul Faculty of Medicine
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qu G, Cui XL, Liu HJ, Ji ZG, Huang YG. Ultrasound-guided Transversus Abdominis Plane Block Improves Postoperative Analgesia and Early Recovery in Patients Undergoing Retroperitoneoscopic Urologic Surgeries: A Randomized Controlled Double-blinded Trial. Chin Med Sci J. 2016 Sep 20;31(3):137-141. doi: 10.1016/s1001-9294(16)30041-4. PMID 27733219
- [Background] Schwarz F, Preusler W, Reifart N, Storger H, Hofmann M, Holscher I. [The long-term success after coronary angioplasty in old age]. Dtsch Med Wochenschr. 1993 Apr 30;118(17):609-14. doi: 10.1055/s-2008-1059369. German. PMID 8482238
- [Background] Copik M, Bialka S, Daszkiewicz A, Misiolek H. Thoracic paravertebral block for postoperative pain management after renal surgery: A randomised controlled trial. Eur J Anaesthesiol. 2017 Sep;34(9):596-601. doi: 10.1097/EJA.0000000000000673. PMID 28731925
- [Background] Parikh BK, Waghmare VT, Shah VR, Mehta T, Butala BP, Parikh GP, Vora KS. The analgesic efficacy of ultrasound-guided transversus abdominis plane block for retroperitoneoscopic donor nephrectomy: A randomized controlled study. Saudi J Anaesth. 2013 Jan;7(1):43-7. doi: 10.4103/1658-354X.109808. PMID 23717232
- See also: Ultrasound-guided Transversus Abdominis Plane Block Improves Postoperative Analgesia and Early Recovery in Patients Undergoing Retroperitoneoscopic Urologic Surgeries: A Randomized Controlled Double-blinded Trial — https://pubmed.ncbi.nlm.nih.gov/27733219/
- See also: Single injection paravertebral block for renal surgery in children — https://pubmed.ncbi.nlm.nih.gov/18482238/
- See also: Thoracic paravertebral block for postoperative pain management after renal surgery A randomised controlled trial — https://pubmed.ncbi.nlm.nih.gov/28731925/
- See also: The analgesic efficacy of ultrasound-guided transversus abdominis plane block for retroperitoneoscopic donor nephrectomy: A randomized controlled study — https://pubmed.ncbi.nlm.nih.gov/23717232/